CLINICAL TRIAL: NCT02139150
Title: Serial FLT PET Imaging in Cancer Patients for Monitoring of Response to Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-050
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Histologically-confirmed Malignancies
Keywords: FLT PET Imaging; 3'deoxy-3' [18F] fluorothymidine ([18F] FLT); CT; scans; 14-050
MeSH Terms: interventions — alovudine; Positron Emission Tomography Computed Tomography

ARMS (1):
- Serial FLT PET Imaging (Experimental): Patients will receive a target injection of up to 10 mCi of FLT. Optionally, dynamic PET imaging over a chosen index lesion (based on size and/or high FDG-avidity on preceding CT and/or FDG PET/CT scans done for clinical purpose such as staging), may be performed. Otherwise, static PET images are obtained at approximately 60 min (+15 min) post FLT injection. In general this "body" scan will cover at least the region from skull base to the upper thigh for extracranial malignancies; depending on the specific location, extremities maybe also be scanned (e.g., extremity sarcoma), or the scan may be restricted to the brain (e.g. glioma).
  Interventions: Radiation: [18F] FLT; Device: PET/CT scans

INTERVENTIONS:
Radiation: [18F] FLT
Device: PET/CT scans

SUMMARY:
The purpose of this study is to see if PET/CT scans that use a radioactive substance called [18F] fluorothymidine (FLT), can detect and monitor changes in the tumor. Radioactive substances are used with PET/CT scans to "see" cancer cells, and are also called radiotracers. FLT is a new radiotracer that has been given to people in prior studies. FLT PET/CT is an experimental scan unlike FDG (fluorodeoxyglucose) PET scan which is a standard clinical scan and is commonly used. The investigators would like to know if there is any evidence of early treatment response by obtaining FLTPET/ CT scans before and after treatment.

DETAILED DESCRIPTION:
This protocol is an "umbrella" or "companion" protocol to be used in conjunction with other protocols that are evaluating treatment response in solid or hematologic malignancies. The aim of this protocol is to determine if PET imaging with the proliferation marker 18FFLT can monitor changes in FLT uptake parameters, in particular changes in the standardized uptake value (SUV), within tumor target lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed (confirmation done at MSKCC) malignancies.
* Patients who have consented to a therapeutic protocol for the treatment of their cancer.
* Patients must be ≥ 18 years old.

Exclusion Criteria:

* Patients who cannot undergo PET/CT scanning (i.e. because of weight limits, claustrophobia).
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
change from pre- to posttreatment | 4 years
  We will describe the distribution of the change and explore if it is associated with the findings of standard-of-care imaging such as FDG-PET or CT/MRI using rank based methods such as Spearman correlation and the signed-ranks test. In addition we will also explore the value of the change in the FLT metrics in predicting the clinical outcome using logistic regression (for response) and proportional hazards regression (for progression and survival).

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/